CLINICAL TRIAL: NCT04680156
Title: An Observational, Double-blind (Sponsor Open), Long-term Study to Evaluate the Safety and Durability (Efficacy) of Response to EN3835 Compared to Placebo in the Treatment of Adhesive Capsulitis of the Shoulder (Frozen Shoulder)
Brief Title: Long-term Follow-up Durability (Efficacy) Study of EN3835 for the Treatment of AC of the Shoulder (Frozen Shoulder)
Status: Terminated | Type: Observational
Why Stopped: Lack of efficacy
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EN3835-223
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EN3835: Previously treated with EN3835 in EN3835-210 or the pivotal phase 3 studies
  Interventions: Drug: Previously treated with EN3835 up to 1.74 mg or Placebo in EN3835-210 or the pivotal phase 3 studies
- Placebo: Previously treated Placebo in EN3835-210 or the pivotal phase 3 studies
  Interventions: Drug: Previously treated with EN3835 up to 1.74 mg or Placebo in EN3835-210 or the pivotal phase 3 studies

INTERVENTIONS:
Drug: Previously treated with EN3835 up to 1.74 mg or Placebo in EN3835-210 or the pivotal phase 3 studies — No treatment to be administered - Observational only

SUMMARY:
This is a long-term follow-up study to evaluate the safety and durability (efficacy) of response to EN3835 compared to placebo in participants who were treated in EN3835-210 or the pivotal Phase 3 parent studies for the treatment of AC of the shoulder (frozen shoulder).

ELIGIBILITY:
Inclusion Criteria:

1. Have been enrolled and completed the EN3835-210 or pivotal Phase 3 parent studies (for Study EN3835-223 eligibility, completed participants are those who were assessed for safety and obtained ASES scores at Day 95/EOS Visit; does not include early terminated participants).
2. Be willing not to use pain medications for the duration of the study period and for 2 weeks prior to the Day 180 visit. Pain medications include but are not limited to: barbiturates, benzodiazepines, methadone, buprenorphine, opioids (e.g., codeine, heroin, hydrocodone, hydromorphone, morphine, oxycodone), and cannabis.

   Note: NSAIDs (ibuprofen, etc.) are allowed.
3. Be willing to undergo MRI of the affected shoulder as required by the protocol.
4. Be able to read, understand, and independently complete patient reported outcome instruments in English.
5. Be willing and able to cooperate with the requirements of the study.
6. Be adequately informed and understand the nature and risks of the study and be able to provide consent.

Exclusion Criteria:

1. Is from a vulnerable population, as defined by the US Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full time, etc.) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the IRB/IEC.
2. Plans to receive (or received prior to Day 180) any invasive or minimally invasive (ie, steroid injections, shoulder manipulation, surgery, etc.) procedures to the affected shoulder during study participation.

   Note: PT is allowed. Any PT received should be captured in the respective electronic case report form (eCRF).
3. Has any contraindications for MRI (implant containing metal, internal metallic object, permanent cosmetics/make-up/tattoos-with exemption of the area to be treated/reviewed, claustrophobia, syncope, low blood pressure, epilepsy, asthma, anemia, or sickle cell disease) as determined by the technologist, the radiologist, and/or investigator performing imaging.
4. Has any other conditions that, in the investigator's opinion, might indicate the participant to be unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants that have completed the EN3835-210 study or the pivotal Phase 3 studies in which they were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Change in ASES composite score in affected shoulder | Days 180, 270, and 360
  The change from Day 95/end of study (EOS) in the parent studies in the adapted American Shoulder and Elbow Society (ASES) composite score for the affected shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kang, Study Director — Endo Pharmaceuticals
Locations (30):
- United States (30):
  - Endo Clinical Trial Site #16, Birmingham, Alabama
  - Endo Clinical Trial Site #9, Mobile, Alabama
  - Endo Clinical Trial Site #25, Tucson, Arizona
  - Endo Clinical Trial Site #8, Encinitas, California
  - Endo Clinical Trial Site #7, Huntington Beach, California
  - Endo Clinical Trial Site #14, La Mesa, California
  - Endo Clinical Trial Site #11, Pasadena, California
  - Endo Clinical Trial Site #2, Clearwater, Florida
  - Endo Clinical Trial Site #19, Fort Lauderdale, Florida
  - Endo Clinical Trial Site #1, Tampa, Florida
  - Endo Clinical Trial Site #4, Winter Park, Florida
  - Endo Clinical Trial Site #26, Dalton, Georgia
  - Endo Clinical Trial Site #20, Lawrenceville, Georgia
  - Endo Clinical Trial Site #21, Newnan, Georgia
  - Endo Clinical Trial Site #24, Stockbridge, Georgia
  - Endo Clinical Trial Site #23, Oak Brook, Illinois
  - Endo Clinical Trial Site #28, Oak Brook, Illinois
  - Endo Clinical Trial Site #10, Stony Brook, New York
  - Endo Clinical Trial Site #29, Durham, North Carolina
  - Endo Clinical Trial Site #13, Dayton, Ohio
  - Endo Clinical Trial Site #30, Altoona, Pennsylvania
  - Endo Clinical Trial Site #12, Indiana, Pennsylvania
  - Endo Clinical Trial Site #5, State College, Pennsylvania
  - Endo Clinical Trial Site #6, Bedford, Texas
  - Endo Clinical Trial Site #17, Bellaire, Texas
  - Endo Clinical Trial Site #27, Georgetown, Texas
  - Endo Clinical Trial Site #22, Laredo, Texas
  - Endo Clinical Trial Site #15, Plano, Texas
  - Endo Clinical Trial Site #18, Plano, Texas
  - Endo Clinical Trial Site #3, Danville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP